CLINICAL TRIAL: NCT06213987
Title: A Control Trial of the Efficacy and Safety of 0.025% Tretinoin Cream and Cream Based in the Treatment of Axillary Hyperpigmentation Associated With Acanthosis Nigricans
Brief Title: The Efficacy Tretinoin Cream in the Treatment of Axillary Hyperpigmentation Associated With Acanthosis Nigricans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Srinakharinwirot University (Other)
Responsible Party: Principal Investigator, Arucha Treesirichod, Associate professor, Srinakharinwirot University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2566URMS0002
Record Dates: First submitted 2023-12-27; First posted 2024-01-19 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Acanthosis Nigricans; Hyperpigmentation
MeSH Terms: conditions — Acanthosis Nigricans; Hyperpigmentation | interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: Intra-individual design with a split-side axillary approach, participants were randomly assigned to apply both 0.025% tretinoin cream and the cream-based product on opposing sides of the axillary region.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: They were allocated the treatment via simple randomization by a third investigator who was not involved in data collection and analysis. Participants were given unlabeled jars of the topical agents. Assessments regarding clinical efficacy will be conducted by an assessor blind to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tretinoin (Experimental): Apply 1 gram of tretinoin cream to the axillary region before bedtime once every other day during the first two weeks, and then once daily after that, total duration of 8 weeks.
  Interventions: Drug: 0.025% Tretinoin
- Cream based (Placebo Comparator): Apply 1 gram of cream based to the axillary region on the opposing side before bedtime once every other day during the first two weeks, and then once daily after that, total duration of 8 weeks.
  Interventions: Drug: 0.025% Tretinoin

INTERVENTIONS:
Drug: 0.025% Tretinoin — Total duration of 8 weeks.

SUMMARY:
The goal of this randomized intra-individual design with a split-side axillary approach is to comparing the efficacy of 0.025% tretinoin cream against a cream-based formulation in the treatment of axillary hyperpigmentation associated with acanthosis nigricans.

The main questions it aims to answer are:

* The efficacy of 0.025% tretinoin cream and cream based in the treatment of axillary hyperpigmentation associated with acanthosis nigricans.
* The safety of 0.025% tretinoin cream and cream based in the treatment of axillary hyperpigmentation associated with acanthosis nigricans.

Participants were randomly assigned to apply both 0.025% tretinoin cream and the cream-based product on opposing sides of the axillary region.

DETAILED DESCRIPTION:
This study employed a randomized intra-individual design with a split-side axillary approach, comparing the efficacy of 0.025% tretinoin cream against a cream-based formulation. Participants were randomly assigned to apply both 0.025% tretinoin cream and the cream-based product on opposing sides of the axillary region. The efficacy of treatment was assessed by Mexameter (melanin index). The investigator's global evaluation (IGE) and parent's global evaluation (PGE) were also used to evaluate the overall success rate. The local safety was conducted for assessment of any cutaneous irritation. At each visit, the investigator graded the degrees of erythema, dryness, peeling, burning, and itching using a scale of 0 to 4. This study was followed for 4 visits, at the baseline, at week 2, 4 and 8.

ELIGIBILITY:
Inclusion Criteria:

* The participants aged over 18 years with BMI more than 25 kg/m2, axillary hyperpigmentation associated with acanthosis nigricans

Exclusion Criteria:

* Vulnerable skin diseases
* Infectious skin diseases
* Other recent diseases involving the axillary
* Other serious medical disorders e.g. liver disease
* Any patients having received other therapies for up to 4 weeks prior to enrollment
* Photosensitive skin
* Immunocompromised host
* Pregnancy and lactation
* Receiving oral retinoids
* Axillary tattoo

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Melanin index assessed by Mexameter | weeks 0, 2, 4 and week 8
  The outcome was treatment efficacy in reducing skin pigmentation, as represented by changes in melanin indices from Mexameter MX18.

SECONDARY OUTCOMES:
Global evaluation scales | weeks 0, 2, 4 and week 8
  The outcomes were improvement in overall assessment using investigator global evaluation scales (IGE) and patient global evaluation scales (PGE), with scores ranging from 0 to 6 (0= clear, 1= almost clear or >90% improvement; 2= marked improvement or >75% improvement; 3= moderate improvement or >50% improvement; 4= mild improvement or >25% improvement; 5= no change; 6= worsening).
Adverse cutaneous reactions | weeks 0, 2, 4 and week 8
  Adverse reactions were explored using the cutaneous irritation grading scales, in which participants rated erythema, dryness, peeling, burning each on a scale of 0 to 4, with 0 representing no adverse effect and 4 as marked severity.

CONTACTS AND LOCATIONS:
Overall Officials: Arucha Treesirichod, Principal Investigator — Srinakharinwirot University
Locations (1):
- Arucha Treesirichod, Ongkharak, Changwat Nakhon Nayok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
In accordance with our commitment to transparency and advancing scientific knowledge, individual participant data collected during this study will be made available for sharing. The data will be accessible to qualified researchers upon request, subject to approval by the data sharing committee.
Supporting Information: Study Protocol
Time Frame: The data release will occur no later than 12 months after the publication of the primary study outcomes.
Access Criteria: Access to the data will be granted based on a set of predefined criteria, and interested parties will be required to submit a formal request outlining the purpose of data usage and plans for analysis. A data sharing agreement may be required to ensure compliance with ethical standards and the protection of participant privacy. For inquiries or to request access to the data, please contact trees_ar@yahoo.com